CLINICAL TRIAL: NCT06290050
Title: A Phase 1, Open-Label, Drug-Drug Interaction Study to Assess the Effect of TAK-279 on the Pharmacokinetics of a Sensitive CYP3A4 Substrate and a Sensitive CYP2C8 Substrate in Healthy Subjects
Brief Title: A Study of the Interaction of Other Drugs With TAK-279 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: TAK-279-1006
Record Dates: First submitted 2024-02-21; First posted 2024-03-04 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — Midazolam; repaglinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A: Midazolam 2 mg (Experimental): Midazolam 2 mg (1 milliliter [mL] of 2 milligram per milliliter [mg/mL]), syrup, orally, on Day 1 of Period 1.
  Interventions: Drug: Midazolam
- Treatment B: Repaglinide 0.5 mg (Experimental): Repaglinide 0.5 mg (1*0.5 mg), tablets, orally, on Day 2 of Period 1.
  Interventions: Drug: Repaglinide
- Treatment C + Treatment A: TAK-279 Dose 1 + Midazolam 2 mg (Experimental): TAK-279 Dose 1, capsules, orally, on Days 1 through 15 of Period 2 followed by Midazolam 2 mg (1 mL of 2 mg/mL), syrup, orally, on Day 14 of Period 2.
  Interventions: Drug: Midazolam; Drug: TAK-279
- Treatment C + Treatment B: TAK-279 Dose 1 + Repaglinide 0.5 mg (Experimental): TAK-279 Dose 1, capsules, orally, on Days 1 through 15 of Period 2 followed by Repaglinide 0.5 mg (1*0.5 mg), tablets, orally, on Day 15 of Period 2.
  Interventions: Drug: Repaglinide; Drug: TAK-279

INTERVENTIONS:
Drug: Midazolam — Midazolam syrup.
  Arms: Treatment A: Midazolam 2 mg; Treatment C + Treatment A: TAK-279 Dose 1 + Midazolam 2 mg
Drug: Repaglinide — Repaglinide tablets.
  Arms: Treatment B: Repaglinide 0.5 mg; Treatment C + Treatment B: TAK-279 Dose 1 + Repaglinide 0.5 mg
Drug: TAK-279 — TAK-279 capsules.
  Arms: Treatment C + Treatment A: TAK-279 Dose 1 + Midazolam 2 mg; Treatment C + Treatment B: TAK-279 Dose 1 + Repaglinide 0.5 mg

SUMMARY:
The main aim of this study is to find out how several doses of TAK-279 affects the body of healthy adults and processes midazolam and repaglinide (pharmacokinetics or PK). Another aim is to learn about the side effects of TAK-279 and how well it is tolerated when given to healthy adults either alone or together with midazolam or repaglinide.

During the study, participants will need to stay at the clinic for 19 days. Blood samples will be taken at several timepoints during the study. The study drug will be given by mouth (orally).

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-279. The study will assess the potential effect of TAK-279 on cytochrome P450 (CYP) 3A4 using the probe substrate midazolam and the potential effect of TAK-279 on CYP2C8 using the probe substrate repaglinide in healthy participants.

The study will enroll approximately 20 participants. Participants will be enrolled in one of the four treatments.

* Treatment A: Midazolam 2 milligram (mg)
* Treatment B: Repaglinide 0.5 mg
* Treatment A + Treatment C: Midazolam 2 mg + TAK-279 Dose 1
* Treatment B + Treatment C: Repaglinide 0.5 mg + TAK-279 Dose 1

This single-center trial will be conducted in the United States. The overall study duration is approximately 59 days including screening period and follow-up.

ELIGIBILITY:
Inclusion Criteria:

Participants must fulfill all of the following inclusion criteria to be eligible for participation in the study:

1. Continuous non-smoker who has not used nicotine and tobacco containing products for at least 3 months prior to the first dosing based on subject self-reporting.
2. Body mass index (BMI) greater than or equal to (>=) 18.0 and less than or equal to (<=) 32.0 kilogram per square meter (kg/m^2) at the screening visit.
3. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, and electrocardiograms (ECGs), as deemed by the investigator or designee, including the following:

   * Seated blood pressure (BP) is >=90/40 millimeter of mercury (mmHg) and <=140/90 mmHg at the screening visit.
   * Seated pulse rate (PR) is >=40 beats per minute (bpm) and <=99 bpm at the screening visit.
   * ECG findings considered normal or not clinically significant by the investigator or designee at the screening visit.
   * Estimated glomerular filtration rate (eGFR) >=80 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) at the screening visit.
   * Liver function tests including Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Alkaline phosphatase (ALP), and total bilirubin <= ULN at the screening visit and at check-in.

Exclusion Criteria:

Participants must not be enrolled in the study if they meet any of the following criteria:

1. Fasting glucose >125 milligram per deciliter (mg/dL) at the screening visit.
2. Has a history or presence of any of the following:

   * Active infection or febrile illness within 7 days prior to first dosing, as assessed by the investigator or designee.
   * Symptoms suggestive of systemic or invasive infection requiring hospitalization or treatment within 8 weeks prior to first dosing.
   * Chronic or recurrent bacterial disease, including but not limited to chronic pyelonephritis or cystitis, chronic bronchitis/pneumonitis, osteomyelitis, or chronic skin ulcerations/infections or fungal infections (except superficial nailbed mycosis).
   * An infected joint prosthesis unless that prosthesis has been removed or replaced greater than 60 days prior to first dosing.
   * Opportunistic infections (example, Pneumocystis jirovecii pneumonia, histoplasmosis, Coccidiomycosis) exception of successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix is not exclusionary.
   * Cancer or lymphoproliferative disease within 5 years prior to first dosing, with the exception of successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix is not exclusionary.
   * Known or suspected condition/illness that is consistent with compromised immunity, including but not limited to any identified congenital or acquired immunodeficiency; splenectomy.
   * Solid organ transplant.
   * Diabetes or prior episode(s) of hypoglycemia.
3. Has history or presence of alcoholism and/or drug abuse within the past 2 years prior to first dosing, as determined by the investigator or designee.
4. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs.
5. History or presence of ventricular dysfunction or risk factors for Torsades de Pointes (example, heart failure, cardiomyopathy, family history of Long QT Syndrome).
6. Positive urine drug or alcohol results at the screening visit or check-in.
7. Unable to refrain from or anticipates the use of:

   * Any drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements including any CYP3A4 and CYP2C8 inhibitors, beginning 14 days prior to the first dosing.
   * Any drugs known to be inducers of CYP3A4 and CYP2C8 enzymes and/or P-gp, including St. John's Wort, for 28 days prior to the first dosing. Appropriate sources (example, Flockhart Table™) including the product label for midazolam and repaglinide will be consulted to confirm lack of PK/pharmacodynamic interaction with the study drugs.
8. Has made a donation of blood or had significant blood loss within 56 days prior to first dosing.
9. Has made a plasma donation within 7 days prior to first dosing.
10. Participated in another clinical study within 30 days prior to first dosing. The 30 day window will be derived from the date of the last dosing in the previous study to Day 1 of Period 1 of the current study.
11. Herpes infections:

    * Has active herpes virus infection, including herpes zoster or herpes simplex 1 and 2 (demonstrated on physical examination and/or medical history) at the screening visit or Day 1 of Period 1.
    * Has history of serious herpetic infection that includes any episode of disseminated disease, multidermatomal herpes zoster virus, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (defined as 2 episodes within 2 years).
12. Positive results for non-herpetic viral diseases at the screening visit:

    * Hepatitis C virus (HCV) antibody and a positive confirmatory test result for HCV Ribonucleic acid (RNA) (nucleic acid test or [Polymerase chain reaction] PCR);
    * Hepatitis B surface antigen (HBsAg+), hepatitis B virus DNA, or Hepatitis B core antibody (HBcAb+) with positive hepatitis B virus Deoxyribonucleic acid (DNA);
    * Human immunodeficiency virus (HIV).
13. Positive results for TB at the screening visit or has the following:

    * Has history of active TB infection, regardless of treatment status.
    * Has signs or symptoms of active TB (including but not limited to chronic fever, chronic productive cough, night sweats, or weight loss) as judged by the investigator or designee.
    * Has evidence of Latent tuberculosis infection (LTBI) as evidenced by a positive QuantiFERON TB Gold (QFT) result OR 2 indeterminant QFT results and does not have documentation of appropriate LTBI prophylaxis. Participants remains eligible if he or she can provide documentation of prior and complete treatment for LTBI (appropriate in duration and type per current local country guidelines).
    * Has had any imaging study prior to the screening visit, including x-ray, chest computed tomography, magnetic resonance imaging, or other chest imaging suggesting evidence of current active or a history of active TB.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for Midazolam and Repaglinide When Administered Alone and With TAK-279 | Period 1-Midazolam Alone: Day 1 predose up to 24 hours (h) postdose; Repaglinide Alone: Day 2 predose up to 16 h postdose; Period 2-Midazolam, With TAK-279: Day 14 predose up to 24 h postdose; Repaglinide with TAK-279:Day 15 predose up to 16 h postdose
AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Midazolam and Repaglinide When Administered Alone and With TAK-279 | Period 1-Midazolam Alone: Day 1 predose up to 24 hours (h) postdose; Repaglinide Alone: Day 2 predose up to 16 h postdose; Period 2-Midazolam, With TAK-279: Day 14 predose up to 24 h postdose; Repaglinide with TAK-279:Day 15 predose up to 16 h postdose
AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Midazolam and Repaglinide When Administered Alone and With TAK-279 | Period 1-Midazolam Alone: Day 1 predose up to 24 hours (h) postdose; Repaglinide Alone: Day 2 predose up to 16 h postdose; Period 2-Midazolam, With TAK-279: Day 14 predose up to 24 h postdose; Repaglinide with TAK-279:Day 15 predose up to 16 h postdose

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) and Adverse Events of Special Interest (AESI) | From Day 1 of Period 1 up to 14 days after the last dose of TAK-279 in Period 2 (up to 29 days)
  An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an AE with an onset that occurs after receiving study drug. AESI (serious or nonserious) includes infections that are severe or serious; opportunistic; herpes virus; active tuberculosis (TB); or any infection requiring intravenous systemic therapy or immunomodulatory therapy, Creatine phosphokinase (CPK) elevation Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 or higher (severe) greater than (>) 5* upper limit of normal (ULN), Liver injury, MACE (Major adverse cardiovascular events), Gastrointestinal perforation, Thromboembolic events, Malignancies including all malignancies, Nonmelanoma skin cancer (NMSC), and excluding NMSC and Lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link — https://clinicaltrials.takeda.com/study-detail/83cee39b850d47a1?idFilter=%5B%22TAK-279-1006%22%5D